CLINICAL TRIAL: NCT02618252
Title: Preventing Delay of Care in Patient With Difficult IV Access: A Randomized Trial of ED Intervention
Brief Title: Ultrasound vs Veinviewer in Patients With Difficulty IV Access
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We were not able to enroll participants
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Quincy Tran, Assosciate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00065438
Record Dates: First submitted 2015-11-04; First posted 2015-12-01 (Estimated); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Vascular Access Complication
Keywords: difficult IV access; ultrasound; veinviewer; near infrared device

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Zonare (Experimental): 108 patients are randomized to receive the intervention of using ultrasound machine (Zonare ZS3 machine) for IV cannulation. These patients will first undergo IV cannulation with assistance of the ultrasound machine.
  Interventions: Device: Zonare
- Veinviewer (Experimental): 108 Patients are randomized to receive the Intervention of using the Veinviewer Flex machine for IV cannulation. These patients will first undergo IV cannulation with assistance of the Veinviewer Flex machine.
  Interventions: Device: Veinviewer

INTERVENTIONS:
Device: Zonare — Patients with difficulty IV access are randomized to receive either intervention with ultrasound machine (Zonare ZS3 machine) or the Veinviewer Flex machine.
  Arms: Zonare
Device: Veinviewer — Patients with difficulty IV access are randomized to receive either intervention with ultrasound machine (Zonare ZS3 machine) or the Veinviewer Flex machine.
  Arms: Veinviewer

SUMMARY:
Patients with difficulty intravenous access frequently have delay of care in emergency departments because Emergency Department (ED) personnel could not establish intravenous (IV) access for diagnostic blood test or treatment. The ultrasound machine or near-infrared devices have been used to improve this situation but no study has ever compared which machine is more efficient. This study is designed to investigate whether the ultrasound or Vein Viewer, which is a near-infrared device, is more efficient.

DETAILED DESCRIPTION:
Intravenous (IV) access is important for patient care in emergency medicine as an estimate of 78% of ED patients would require more than 3 ED resources such as blood tests, medication, contrast, fluid. Care for patients with difficult intravenous access (DIVA) could be significantly delayed as it may take up to 120 minutes to establish IV access in patients with severe DIVA. Many solutions for DIVA had also been established to avoid central venous catheter insertion, including using ultrasound or near-infrared imaging systems for peripheral IV insertion.

Using ultrasound in the ED has been shown to decrease the rate of central venous catheters (CVC) insertion. However, the results from ultrasound-guided peripheral IV insertion (USGPIV) have been mixed. Among patients with DIVA, Costantino reported USGPIV required less time to successful first cannulation and fewer punctures comparing to traditional approach of landmark and palpation. However, other studies showed that USGPIV did not improve successful first attempts comparing to traditional IV insertion, and may have taken same or even longer time to successfully establish IV. USGPIV success rate requires more training for nurses and ED technicians as it is operator - dependent.

Patients have difficulty with IV access because their veins' clinical accessibility is low, for example, they are less visible or less palpable. The near-infrared imaging devices, such as Christie Digital's VeinViewer, improve this situation by using infra-red lights to make veins visible to the eyes.

Compared with routine IV insertion, near-Infra red imaging devices have been shown to increase first successful attempts and in less time in children with DIVA and improved visualization of peripheral veins. However, it did not show higher rate of successful attempts nor faster time in non-selected adults.

The efficacy of these near-infrared devices has not been established among adult patients with DIVA.

ELIGIBILITY:
Inclusion Criteria:

* Patients who fail inspections for visible or palpable veins or
* Patients who request Ultrasound guided peripheral IV (USGPIV)
* patients who are oriented to self (correct last name, first name), place (correct name of hospital), time (correct day of week or month of year) and person (correct name of current president)

Exclusion Criteria:

* Patients < 18 years of age
* Patients with hemodynamically instability requiring rapid central access.
* Patients with impaired cognition and not able to consent, these patients are :

  * Clinically intoxicated patients, as defined by primary team.
  * Patients who family reported as "confused", "confusion", "altered mental status."
  * Patients who is not oriented x 4 as above
* Patients who do not speak English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Operator's time | up to 40 minutes
  time from equipment-in-room to successful aspiration of 3ml of blood

SECONDARY OUTCOMES:
Number of first successful attempts | 40 minutes
  operators have up to 40 minutes or 3 attempts.
Number of failures | 40 minutes
  operators have up to 40 minutes or 3 attempts prior to patients crossing over or requiring a rescue modality
IV size | 40 minutes
  operators have up to 40 minutes or 3 attempts to establish IV from 18 to 24 gauge
Patient satisfaction | up to 40 minutes
  after completion of IV cannulation
Patient's perception of pain | up to 40 minutes
  after completion of IV cannulation
ED length of stay | 24 hours
  Length of stay for discharged patients.
hospital length of stay for admitted patient | 30 days
  Length of stay for admitted patients
Cannulation time | 40 minutes
  time from applying tourniquet to successful aspiration of 3ml of blood.
Number of failure to cannulate | 40 minutes
  operators have up to 40 minutes or 3 attempts.

CONTACTS AND LOCATIONS:
Overall Officials: Quincy Tran, MD, PhD, Principal Investigator — University of Maryland
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tanabe P, Gimbel R, Yarnold PR, Adams JG. The Emergency Severity Index (version 3) 5-level triage system scores predict ED resource consumption. J Emerg Nurs. 2004 Feb;30(1):22-9. doi: 10.1016/j.jen.2003.11.004. PMID 14765078
- [Background] Witting MD. IV access difficulty: incidence and delays in an urban emergency department. J Emerg Med. 2012 Apr;42(4):483-7. doi: 10.1016/j.jemermed.2011.07.030. Epub 2011 Dec 2. PMID 22137793
- [Background] Bauman M, Braude D, Crandall C. Ultrasound-guidance vs. standard technique in difficult vascular access patients by ED technicians. Am J Emerg Med. 2009 Feb;27(2):135-40. doi: 10.1016/j.ajem.2008.02.005. PMID 19371518
- [Background] Maiocco G, Coole C. Use of ultrasound guidance for peripheral intravenous placement in difficult-to-access patients: advancing practice with evidence. J Nurs Care Qual. 2012 Jan-Mar;27(1):51-5. doi: 10.1097/NCQ.0b013e31822b4537. PMID 21826027
- [Background] Teismann NA, Knight RS, Rehrer M, Shah S, Nagdev A, Stone M. The ultrasound-guided "peripheral IJ": internal jugular vein catheterization using a standard intravenous catheter. J Emerg Med. 2013 Jan;44(1):150-4. doi: 10.1016/j.jemermed.2012.02.044. Epub 2012 May 11. PMID 22579025
- [Background] Weiner SG, Sarff AR, Esener DE, Shroff SD, Budhram GR, Switkowski KM, Mostofi MB, Barus RW, Coute RA, Darvish AH. Single-operator ultrasound-guided intravenous line placement by emergency nurses reduces the need for physician intervention in patients with difficult-to-establish intravenous access. J Emerg Med. 2013 Mar;44(3):653-60. doi: 10.1016/j.jemermed.2012.08.021. Epub 2012 Oct 25. PMID 23103067
- [Background] de Graaff JC, Cuper NJ, Mungra RA, Vlaardingerbroek K, Numan SC, Kalkman CJ. Near-infrared light to aid peripheral intravenous cannulation in children: a cluster randomised clinical trial of three devices. Anaesthesia. 2013 Aug;68(8):835-45. doi: 10.1111/anae.12294. Epub 2013 Jun 14. PMID 23763614
- [Background] Shokoohi H, Boniface K, McCarthy M, Khedir Al-tiae T, Sattarian M, Ding R, Liu YT, Pourmand A, Schoenfeld E, Scott J, Shesser R, Yadav K. Ultrasound-guided peripheral intravenous access program is associated with a marked reduction in central venous catheter use in noncritically ill emergency department patients. Ann Emerg Med. 2013 Feb;61(2):198-203. doi: 10.1016/j.annemergmed.2012.09.016. Epub 2012 Nov 7. PMID 23141920
- [Background] Au AK, Rotte MJ, Grzybowski RJ, Ku BS, Fields JM. Decrease in central venous catheter placement due to use of ultrasound guidance for peripheral intravenous catheters. Am J Emerg Med. 2012 Nov;30(9):1950-4. doi: 10.1016/j.ajem.2012.04.016. Epub 2012 Jul 15. PMID 22795988
- [Background] Costantino TG, Parikh AK, Satz WA, Fojtik JP. Ultrasonography-guided peripheral intravenous access versus traditional approaches in patients with difficult intravenous access. Ann Emerg Med. 2005 Nov;46(5):456-61. doi: 10.1016/j.annemergmed.2004.12.026. PMID 16271677
- [Background] Stein J, George B, River G, Hebig A, McDermott D. Ultrasonographically guided peripheral intravenous cannulation in emergency department patients with difficult intravenous access: a randomized trial. Ann Emerg Med. 2009 Jul;54(1):33-40. doi: 10.1016/j.annemergmed.2008.07.048. Epub 2008 Sep 27. PMID 18824276
- [Background] Liu YT, Alsaawi A, Bjornsson HM. Ultrasound-guided peripheral venous access: a systematic review of randomized-controlled trials. Eur J Emerg Med. 2014 Feb;21(1):18-23. doi: 10.1097/MEJ.0b013e328363bebc. PMID 23880981
- [Background] Witting MD, Schenkel SM, Lawner BJ, Euerle BD. Effects of vein width and depth on ultrasound-guided peripheral intravenous success rates. J Emerg Med. 2010 Jul;39(1):70-5. doi: 10.1016/j.jemermed.2009.01.003. Epub 2009 Mar 9. PMID 19272730
- [Background] Sebbane M, Claret PG, Lefebvre S, Mercier G, Rubenovitch J, Jreige R, Eledjam JJ, de La Coussaye JE. Predicting peripheral venous access difficulty in the emergency department using body mass index and a clinical evaluation of venous accessibility. J Emerg Med. 2013 Feb;44(2):299-305. doi: 10.1016/j.jemermed.2012.07.051. Epub 2012 Sep 13. PMID 22981661
- [Background] Hess HA. A biomedical device to improve pediatric vascular access success. Pediatr Nurs. 2010 Sep-Oct;36(5):259-63. PMID 21067078
- [Background] Kim MJ, Park JM, Rhee N, Je SM, Hong SH, Lee YM, Chung SP, Kim SH. Efficacy of VeinViewer in pediatric peripheral intravenous access: a randomized controlled trial. Eur J Pediatr. 2012 Jul;171(7):1121-5. doi: 10.1007/s00431-012-1713-9. Epub 2012 Mar 14. PMID 22415409
- [Background] Sun CY, Lee KC, Lin IH, Wu CL, Huang HP, Lin YY, Hsu YF, Yu HR. Near-infrared light device can improve intravenous cannulation in critically ill children. Pediatr Neonatol. 2013 Jun;54(3):194-7. doi: 10.1016/j.pedneo.2012.12.012. Epub 2013 Feb 1. PMID 23597539
- [Background] Aulagnier J, Hoc C, Mathieu E, Dreyfus JF, Fischler M, Le Guen M. Efficacy of AccuVein to facilitate peripheral intravenous placement in adults presenting to an emergency department: a randomized clinical trial. Acad Emerg Med. 2014 Aug;21(8):858-63. doi: 10.1111/acem.12437. PMID 25176152
- [Background] Fields JM, Piela NE, Au AK, Ku BS. Risk factors associated with difficult venous access in adult ED patients. Am J Emerg Med. 2014 Oct;32(10):1179-82. doi: 10.1016/j.ajem.2014.07.008. Epub 2014 Jul 30. PMID 25171796